CLINICAL TRIAL: NCT03899012
Title: Validation of the Data Quality of the EVEREG Incisional Hernia Surgery Registry
Brief Title: Audit of the EVEREG Incisional Hernia Registry (AUDHIT)
Acronym: AUDHIT
Status: Completed | Type: Observational
Sponsor: Hospital Universitari Joan XXIII de Tarragona. (Other)
Responsible Party: Principal Investigator, Carles Olona Casas, Consultant General and Digestive Surgeon, Hospital Universitari Joan XXIII de Tarragona.
Other Study IDs: AUDHIT
Record Dates: First submitted 2019-03-29; First posted 2019-04-02 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Incisional Hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Incisional Hernia Surgery — Verification of the accuracy in the collection of 21 selected variables in the Spanish EVEREG Incisional Hernia Surgery Registry

SUMMARY:
Objective: The objective of the study is to verify and validate the data collected in the EVEREG Incisional Hernia Surgery Registry between 2012 and 2018 through an audit process.

Methods: An audit of registered cases (Incisional Hernia Patients undergoing surgery) from 2012 to 2018, and a descriptive analysis of these data will be performed Expected results: The study could show that the EVEREG Incisional Hernia Registry is a reliable source of information, valid for carrying out specific and exhaustive analysis that may lead to high quality publications.

Relevance: The standardization of the data collection is very important to compare outcomes between different centers. This study will allow us to verify the accuracy of the collected data

DETAILED DESCRIPTION:
Objective: The objective of the study is to verify and validate the data collected in the EVEREG Incisional Hernia Surgery Registry between 2012 and 2018 through an audit process Secondary objective are a descriptive analysis of the registered data and a comparison with the outcomes published in other studies

Background The high volume of data obtained by well-validated registries allows them to be considered appropriate for the study of their multiple variables, even when the differences are small and the variables are rare.

The use of registries of abdominal wall surgery has been extended in recent years worldwide and the analysis of their data has already improved the knowledge and treatment of this pathology of high prevalence. The National Registry of Incisional Hernia (EVEREG), is promoted by the Section of Abdominal Wall and Sutures of the Spanish Association of Surgeons, collecting the data prospectively. It began in July 2012. In December 2018 it included data from 160 Spanish hospitals, and a total of 9780 cases of incisional hernias. Hernias related to a previous laparotomy are included, primary ventral hernias are not recorded, and the first analyzes have already been published.

The validity of any registry is based on the accuracy of the data. For this reason, it is considered very important to perform the audit in the centers where the data have been recorded in the EVEREG on-line registry.

METHODOLOGY

Population to study The data of all the patients included in the EVEREG Incisional Hernia registry will be compiled and analyzed from July 2012 to December 2018.

Once the approval by the corresponding Ethics Committee has been obtained, audits will be carried out in each center. A group of 2 researchers from a center different from the one evaluated, will carry out an exhaustive review of the variables previously determined and collected in the registry. The reviewers will prepare an audit report, previously designed by the PIs, where the results obtained for each variable studied will be collected. In the last 3 months of the study the statistical analysis and writing of conclusions will be carried out Study variables The EVEREG registry includes 68 patient parameters divided into sections corresponding to: patient history , characteristics of the incisional hernia , characteristics of the intervention and complications and follow-up of the patient up to 2 years postoperatively They are open variables and agreed by consensus of the group, updates have been made with the aim of their improvement. Due to the different number of cases introduced per center and in order to obtain a sufficiently representative sample of the total number of cases introduced and of the various variables under study, the selection of the sample has been designed taking into account the total number of cases to be selected and a minimum of cases of each center to avoid the standard error and the sampling error.

A selection of the variables to be analyzed was made according to their clinical relevance:

* Personal Background: Age, Size, Weight
* Incisional hernia: Type, Trocar, Paraestomal, Pneumoperitoneum preop, Botulinum toxin
* Intervention: Date, Access, Components Separation, Mesh Placement, Mesh Number, Mesh Type, Mesh Position, Complications, High
* Postoperative 1: Date, Complications
* Last Postoperative Control: Date, Complications

Statistical analysis plan Univariate descriptive analysis will be performed, presenting the results as means (with standard deviation and range) for the continuous variables and as numbers and percentages for the categorical variables. In addition, bivariate analysis will be carried out among the variables of interest to describe their level of correlation and evaluate the possible differences between them. To evaluate the differences between the continuous variables, the comparison of means based on the T-Student will be used, and for the comparison of differences in the categorical variables, the Chi-square test will be used. Finally, linear regression models and generalized linear models (as appropriate depending on the response variable) will be used to study the dependence of the variables of interest, with other factors of study. Statistical analysis will be carried out using the SPSS (Statistical Package for the Social Sciences) Software (IBM SPSS Statistics 22). All tests will be bilateral with a level of significance of 5%. 100% of the data recorded from 01/01/2014 to 06/30/2017 will be analyzed, and the proportion of values lost in the variables of interest will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* data of all the patients treated in the Hospitals of Catalonia and included in the EVEREG registry of Hernia Incisional from July 2012 to December 2018

Exclusion Criteria:

* Patients not registered previously in the EVEREG registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The data of all the patients treated in the Hospitals of Catalonia and included in the EVEREG registry of Hernia Incisional from July 2012 to December 2018 will be compiled and analyzed.
Sampling Method: Probability Sample
Enrollment: 337 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2022-02-15 (Actual)

PRIMARY OUTCOMES:
Data accuracy | 2 Years
  Determining the case ascertainment percentage for the Spanish EVEREG Incisional Hernia Surgery Registry

CONTACTS AND LOCATIONS:
Overall Officials: Carles Olona, PhD, Principal Investigator — Consultant General and Digestive Surgeon
Locations (1):
- Hospital Universitari de Tarragona Joan XXIII, Tarragona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Olona C, Pereira-Rodriguez JA, Comas J, Villalobos R, Alonso V, Amador S, Bombuy E, Mitru C, Gimeno M, Lopez-Cano M. Data quality validation of the Spanish Incisional Hernia Surgery Registry (EVEREG): pilot study. Hernia. 2023 Jun;27(3):665-670. doi: 10.1007/s10029-023-02782-3. Epub 2023 Mar 24. PMID 36964455